CLINICAL TRIAL: NCT04979923
Title: Efficacy of Nebulized Lidocaine, Salbutamol, and Beclomethasone Plus Salbutamol in the Covid-19 Patients With ARDS on Non-invasive Ventilation; Randomized Control Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Sairah Sadaf, Associate Professor, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 227/IRB/SZMC/SZH
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine group (Experimental)
  Interventions: Drug: Lidocaine
- Salbutamol group (Placebo Comparator)
  Interventions: Drug: Lidocaine
- Beclomethasone plus salbutamol (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine will be used for nebulization of the covid-19 patients and will be compared with other two drugs

SUMMARY:
The COVID-19, a pandemic as declare by WHO1, has a devastating impact on health and economic worldwide2. Literature suggests that acute respiratory distress syndrome (ARDS) develops over 20% of the infected individuals with Coivd-pneumonia3 along with other symptoms like fever followed by cough and dyspnea as well as chest pain in severe cases4. The current preventative strategies are non-specific10, and current interventions are predominantly supportive1. Recently, some studies have demonstrated anti-inflammatory actions for local anesthetics including lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 positive
* Moderate to severe ARDS

Exclusion Criteria:

* patients with COPD or taking bronchodilators and steroids for chronic respiratory illnesses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Cough suppression | within five minutes of initiation of treatment it will be assessed
  it will be assessed by using cough severity score

SECONDARY OUTCOMES:
correction of hypoxia | immediately before and after intervention
  it will be assessed by PaO2

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed medical college & hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided